CLINICAL TRIAL: NCT04441515
Title: Music After Stroke To Enhance Rehabilitation
Acronym: MASTER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pace University (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MASTER1
Record Dates: First submitted 2020-06-10; First posted 2020-06-22 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Stroke, Acute; Expressive Aphasia; Movement, Abnormal; Depressive Disorder
MeSH Terms: conditions — Stroke; Aphasia, Broca; Dyskinesias; Depressive Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music (Experimental): music supplied by ipod
  Interventions: Device: Ipod with music
- oral books (Active Comparator): Listening to books on ipod
  Interventions: Device: ipod with books to listen
- usual care (Placebo Comparator): Usual care
  Interventions: Device: ipod only with usual care

INTERVENTIONS:
Device: Ipod with music — music of patient's preference provided 2 hours daily
  Arms: Music
Device: ipod with books to listen — 2 hours of daily listening to books
  Arms: oral books
Device: ipod only with usual care — participants given device only
  Arms: usual care

SUMMARY:
Music that is familiar and preferred by patients has been shown to heighten neuroplasticity and can mitigate these disabilities. Therefore, this study seeks to explore the effect of providing patient preferred music to patients in the very early post stroke period (within 24 hours of a left cerebral artery stroke [LMCA]event) as a complementary modality to usual stroke care.

DETAILED DESCRIPTION:
Aim I. The primary aim of MASTER is to identify whether a potential relationship exists between an intervention of participant preferred music, when initiated within the first 24 hours following a left middle cerebral artery stroke, and a reduction in the following disabilities: Expressive aphasia, right hand functional deficit and post stroke depression. This aim will serve to address the first research hypothesis and address the relationship between These disabilities are well known sequalae among patients diagnosed with the most common form of stroke, a LMCA stroke. Participant preferred music within the first 24 hours following a LMCA stroke and a reduction in: Expressive aphasia, right hand functional deficit and post stroke depression, as these disabilities are well known sequalae among LMCA stroke patients.

Aim II. The second aim of MASTER is to identify if a relationship exists between an intervention of audible books, when initiated within the first 24 hours following a LMCA stroke, and a reduction in the following disabilities: Expressive aphasia, right hand functional deficit and post stroke depression.

Sufficient evidence exists to suggest that although listening to books stimulates cognitive function, the effect of melody and participant engagement in music is far superior to listening to words alone as the inherent rhythmicity of patient-favored music has been shown to strengthen synchronous neuronal connectivity, by modulating dopamine and inducing fine grained neuroanatomical changes in a recovering brain.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of LMCA stroke within prior 24 hours
* Not identified as critically ill
* Glascow Coma Scale > 8 at time of consent
* Resident of a home with a land line or cell phone
* Able to speak in English or Spanish prior to stroke event
* Presence of expressive aphasia at time of enrollment.

Exclusion Criteria:

* Stroke diagnosis other than LMCA territory stroke
* Unable to provide consent by patient or legally accountable person acting on behalf of the patient (healthcare proxy, healthcare power of attorney), Patient/ representative
* Does not speak English or Spanish prior to stroke event
* Have a diagnosis of end stage cancer, or other medical conditions that dramatically increase a risk of mortality within one year
* Any pre-existing communication disorder (including dementia)
* Patients that are deemed critically ill will not be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-04-30 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
expressive aphasia measured by use of the WAB-R | 6 months
  Change in expressive aphasia will be measured by use of the WAB-R. Western Aphasia Battery-Revised (WAB- R).This instrument is intended to provide a standardized measure of aphasia type and severity. Implementation of the instrument takes 15 approximately minutes to complete. THE WAB-R identifies and classifies 8 aphasia types: Global, Broca's, Isolation, Transcortical Motor, Wernicke's, transcortical Sensory, Conduction and Anomic. The WAB-R assesses linguistic skills more frequently affected by aphasia. Participants will be assessed at enrollment, discharge from hospital and again at 1,3,6 months post stroke.
motor activity right hand as measured using the Motor Activity log | 6 months
  Change in right hand motor activity and function will be assessed using the Motor Activity Log. The Motor Activity Log (MAL) is a semi-structured interview for hemiparetic stroke patients to assess the use of their paretic arm and hand Target tasks include object manipulation (e.g. pen, fork, comb, and cup) as well as the use of the arm during gross motor activities (e.g. transferring to a car, steadying oneself during standing, pulling a chair into a table while sitting). Participants will be assessed at enrollment, discharge from hospital and again at 1,3,6 months post stroke.
Depressive symptoms as measured using the PHQ-9 | 6 months
  A change in depressive symptoms will be assessed using the PHQ-9. The PHQ-9 will be used for screening for depression, as it has been identified as the preferred (gold standard) screening tool for depression among post stroke patients in hospitals. The PHQ-9 takes less than 5 minutes to administer, and has been shown to have superior sensitivity and specificity.
Quality of life as measured using the 20 item short form survey (SF-20) | 6 months
  Change quality of life is assessed in this study, a 20-item short form survey (SF-20) will be used to assess quality of life. Participants will be assessed at enrollment, discharge from hospital and again at 1,3,6 months post stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Millie Hepburn, PhD, Principal Investigator — Pace University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flanagan J. (1978). A research approach to improving our quality of life. American Psychologist, 33, 138-147.
- [Background] Kertesz, A. (2006). Western Aphasia Battery-Revised. San Antonio, TX: Pearson.
- [Result] Amengual JL, Rojo N, Veciana de Las Heras M, Marco-Pallares J, Grau-Sanchez J, Schneider S, Vaquero L, Juncadella M, Montero J, Mohammadi B, Rubio F, Rueda N, Duarte E, Grau C, Altenmuller E, Munte TF, Rodriguez-Fornells A. Sensorimotor plasticity after music-supported therapy in chronic stroke patients revealed by transcranial magnetic stimulation. PLoS One. 2013 Apr 17;8(4):e61883. doi: 10.1371/journal.pone.0061883. Print 2013. PMID 23613966
- [Result] Carver DJ, Chapman CA, Thomas VS, Stadnyk KJ, Rockwood K. Validity and reliability of the Medical Outcomes Study Short Form-20 questionnaire as a measure of quality of life in elderly people living at home. Age Ageing. 1999 Mar;28(2):169-74. doi: 10.1093/ageing/28.2.169. PMID 10350414
- [Result] Edmonds LA, Donovan NJ. Item-level psychometrics and predictors of performance for Spanish/English bilingual speakers on an object and action naming battery. J Speech Lang Hear Res. 2012 Apr;55(2):359-81. doi: 10.1044/1092-4388(2011/10-0307). Epub 2012 Jan 3. PMID 22215032
- [Result] Fox K, Stryker M. Integrating Hebbian and homeostatic plasticity: introduction. Philos Trans R Soc Lond B Biol Sci. 2017 Mar 5;372(1715):20160413. doi: 10.1098/rstb.2016.0413. PMID 28093560
- [Result] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Result] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL; American Heart Association Stroke Council. 2018 Guidelines for the Early Management of Patients With Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2018 Mar;49(3):e46-e110. doi: 10.1161/STR.0000000000000158. Epub 2018 Jan 24. PMID 29367334
- [Result] Kim M, Tomaino CM. Protocol evaluation for effective music therapy for persons with nonfluent aphasia. Top Stroke Rehabil. 2008 Nov-Dec;15(6):555-69. doi: 10.1310/tsr1506-555. PMID 19158063
- [Result] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Result] Scholz DS, Rohde S, Nikmaram N, Bruckner HP, Grossbach M, Rollnik JD, Altenmuller EO. Sonification of Arm Movements in Stroke Rehabilitation - A Novel Approach in Neurologic Music Therapy. Front Neurol. 2016 Jun 30;7:106. doi: 10.3389/fneur.2016.00106. eCollection 2016. PMID 27445970
- [Result] Uswatte G, Taub E, Morris D, Light K, Thompson PA. The Motor Activity Log-28: assessing daily use of the hemiparetic arm after stroke. Neurology. 2006 Oct 10;67(7):1189-94. doi: 10.1212/01.wnl.0000238164.90657.c2. PMID 17030751
- [Result] van der Lee JH, Beckerman H, Knol DL, de Vet HC, Bouter LM. Clinimetric properties of the motor activity log for the assessment of arm use in hemiparetic patients. Stroke. 2004 Jun;35(6):1410-4. doi: 10.1161/01.STR.0000126900.24964.7e. Epub 2004 Apr 15. PMID 15087552